CLINICAL TRIAL: NCT07332234
Title: Utility of Optic Nerve Ultrasonography in Assessing Cerebral Inflammation and Intracranial Hypertension in Patients With Cerebral Impairment
Brief Title: Optic Nerve Ultrasound for Assessing Cerebral Inflammation and Intracranial Hypertension in Cerebral Pathologies
Acronym: EICON
Status: Recruiting | Type: Observational
Sponsor: Spitalul Clinic de Boli Infecțioase și tropicale "Dr. Victor Babeș" (Other)
Collaborators: Institutul Clinic Fundeni (Other)
Responsible Party: Principal Investigator, Bogdan Pavel, MD, PhD, DESA, Spitalul Clinic de Boli Infecțioase și tropicale "Dr. Victor Babeș"
Other Study IDs: 18261-14/10/2025
Record Dates: First submitted 2025-12-03; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Meningitis; Meningitis/Encephalitis; Stroke; Ultrasound; Intracranial Hypertension; Cerebral Tumors
Keywords: ONSD; Optic Nerve Sheath Diameter; Intracranial hypertension; Meningitis; Encephalitis; Stroke; Cerebral tumors
MeSH Terms: conditions — Meningitis; Encephalitis; Stroke; Intracranial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Infectious Pathology Group: Patients admitted into the hospital with suspected meningitis or encephalitis
  Interventions: Diagnostic Test: Optic Nerve Sheath Diameter
- Non-Infectious Pathology Group: Patients admitted into the hospital with suspected stroke or cerebral tumors (non-infectious pathology)
  Interventions: Diagnostic Test: Optic Nerve Sheath Diameter

INTERVENTIONS:
Diagnostic Test: Optic Nerve Sheath Diameter — Ultrasonographic measurement of the optic nerve sheath diameter
  Other Names: Ocular Ultrasound; Optic Nerve Sheath Ultrasonographic Diameter

SUMMARY:
Timely detection of signs of raised intracranial pressure or persistent inflammation within the meninges can expedite therapeutic decisions improving the prognosis of patients with brain damage. Optic nerve ultrasonography provides a user-friendly, safe, low-cost, and non-invasive imaging method that can be easily deployed for ICU patient assessment. This study aims to evaluate the sensitivity and specificity of optic nerve ultrasound in estimating cerebral inflammation extension and cerebral edema in patients in the ICU. The working hypothesis is that optic nerve ultrasound is a useful tool in the rapid diagnosis of cerebral edema and the presence or persistence of cerebral inflammation, which can enable adapted and rapid therapeutic interventions.

DETAILED DESCRIPTION:
"Utility of Optic Nerve Ultrasonography in Assessing Cerebral Inflammation and Intracranial Hypertension in Patients with Cerebral Impairment" - briefly, the EICON Study.

Investigators Principal Investigator (1): Bogdan PAVEL, MD, PhD, DESA, "Dr. Victor Babes" Clinical Hospital of Infectious and Tropical Diseases.

Principal Investigator (2): Sebastian ISAC, MD, PhD, DESA, Fundeni Clinical Institute Principal Investigator (3): Prof. Gabriela DROC, M.D., Ph.D., Fundeni Clinical Institute

Study Design Study Type: Observational Estimated Number of Participants: 200 participants Primary Purpose: Evaluation Actual Study Start Date: December 1st, 2025 Estimated Primary Completion Date: December 1st, 2027 Estimated Study Completion Date: December 1st, 2027

Groups and Interventions

Group 1: Infectious Pathology Group

Patients admitted with suspected meningitis or encephalitis will undergo the following investigations:

Assessment of consciousness using validated scales (GCS, RASS).

Optic nerve ultrasound to measure the optic nerve sheath diameter (ONSD), performed according to the following protocol:

The patient is positioned supine at a 20-30° incline. A linear probe (9-10 MHz; depth=40 mm; focus=30 mm) is used. The optic nerve must be visible at least 6 mm posterior to the retina. The retinal artery is identified. The diameter of the optic nerve is measured 3 mm posterior to the retina in both the transverse and sagittal planes; the reported value is the mean of the two measurements.

Measurements are performed independently by two examiners. Transcranial Doppler (TCD) to determine the pulsatility index of the middle cerebral artery.

Computed tomography (CT) to exclude intracranial hypertension. Lumbar puncture with measurement of cerebrospinal fluid (CSF) opening pressure. Blood sampling for C-reactive protein (CRP) and neuron-specific enolase (NSE) levels.

Daily Monitoring During Hospitalization:

Daily assessment of consciousness (GCS, RASS) at 09:00. Daily optic nerve ultrasound at 09:00 following the protocol described above. Daily TCD examination of the middle cerebral artery at 09:10. CT scan if clinical signs of intracranial hypertension develop or if there is a sudden decline in GCS of >3 points.

Repeat lumbar puncture with CSF pressure measurement at 72 hours and 7 days after admission.

Blood sampling for CRP, NSE, and total antioxidant capacity at admission, 72 hours, and 7 days.

Group 2: Patients With Non-Infectious Neurological Pathology

Patients admitted with suspected stroke (CVA), brain tumors, or metabolic encephalopathy will undergo the following investigations:

Assessment of consciousness using validated scales (GCS, RASS).

Optic nerve ultrasound to measure the optic nerve sheath diameter (ONSD), performed according to the following protocol:

The patient is positioned supine at a 20-30° incline. A linear probe (9-10 MHz; depth=40 mm; focus=30 mm) is used. The optic nerve must be visible at least 6 mm posterior to the retina. The retinal artery is identified. The diameter of the optic nerve is measured 3 mm posterior to the retina in both the transverse and sagittal planes; the reported value is the mean of the two measurements.

Measurements are performed independently by two examiners. Transcranial Doppler (TCD) to determine the pulsatility index of the middle cerebral artery.

Computed tomography (CT) to exclude intracranial hypertension. Lumbar puncture with measurement of cerebrospinal fluid (CSF) opening pressure. Blood sampling for C-reactive protein (CRP) and neuron-specific enolase (NSE) levels.

Daily Monitoring During Hospitalization:

Daily assessment of consciousness (GCS, RASS) at 09:00. Daily optic nerve ultrasound at 09:00 following the standardized measurement protocol.

Daily TCD examination at 09:10 to assess the middle cerebral artery pulsatility index.

CT scan if signs of intracranial hypertension appear or if the GCS decreases abruptly by >3 points.

Lumbar puncture with CSF pressure measurement at 72 hours and 7 days after admission (if applicable).

Blood sampling for CRP and NSE levels at 72 hours and 7 days after admission.

General Objectives

1. Primary Objectives:

   To evaluate the sensitivity and specificity of optic nerve ultrasound in the assessment of cerebral inflammation and cerebral edema.

   To establish threshold values for diagnosing intracranial hypertension, according to the specific pathology.

   To correlate the optic nerve diameter with the patients' clinical condition.
2. Secondary Objectives:

28-day mortality Quality of life assessment on day 28 Rate of local and systemic complications

Inclusion Criteria:

* Patients admitted into one of the specified wards of the involved hospitals
* Patients aged 18-60 years
* Suspected meningitis, encephalitis, stroke or cerebral tumors

Exclusion Criteria:

* Age under 18 years or over 60 years old
* Ocular lesions preventing ocular ultrasound (palpebral infections, cornean erosions, glaucoma, trauma)
* Conditions preventing lumbar puncture (coagulation disorders, epidural abscesses, local infections)

All data is collected and stored electronically, using a tabular Excel file shared by all investigators.

Ethical Considerations: For this study, we request deferred consent and invoke the emergency consent procedure for medical research, in accordance with Article 6, paragraph 4 of the WMO. This approach is justified for the following reasons:

Patients admitted to infectious disease, neurology, or intensive care units often lack the capacity to provide informed consent. Under the Medical Treatment Act (WGBO), individuals who may serve as legal representatives include: a pre-designated representative, a spouse, a registered or other life partner, a parent or child, a sibling, and, in some cases, a court-appointed guardian. However, legal representatives are frequently not present when patients are admitted to the ICU or when the inclusion criteria are met. Moreover, obtaining informed consent from a legal representative requires sufficient time for them to review and consider the information provided. In the acute phase of admission-particularly in the ICU-legal representatives are naturally focused on the patient's clinical status rather than participation in research.

Procedures for Obtaining Consent Informed consent will be requested from the legal representative as soon as possible and no later than 48 hours after the inclusion criteria are met. If feasible, informed consent will be obtained in advance.

If informed consent from the legal representative is not obtained within 48 hours, or if the representative refuses participation within this period, the patient will be excluded and all collected data will be removed from the study.

The legal representative will receive both oral and written information, provided either in person or via telephone and email. Written informed consent may be returned by email within 12 hours of receiving the information, but always within the 48-hour window following inclusion.

Consent received by email must subsequently be confirmed with a signed paper form as soon as possible, and no later than 48 hours after the emailed confirmation.

Retrospective Consent From the Patient A second informed consent procedure will be conducted retrospectively once the patient regains capacity and is able to adequately understand the situation. At that time, the study information will be provided directly to the patient, and written informed consent will be requested and signed by both the patient and the executive investigator. If the patient declines participation, all data collected up to that point will be permanently deleted.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted into one of the specified wards of the involved hospitals
* Patients aged 18-60 years
* Suspected meningitis, encephalitis, stroke or cerebral tumors

Exclusion Criteria:

* Age under 18 years or over 60 years old
* Ocular lesions preventing ocular ultrasound (palpebral infections, cornean erosions, glaucoma, trauma)
* Conditions preventing lumbar puncture (coagulation disorders, epidural abscesses, local infections)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients admitted into the Anesthesia and Intensive Care Department of the Fundeni Clinical Institute in Bucharest, and the Anesthesia and Intensive Care Department and Infectious Diseases departments of the "Dr. Victor Babes" Hospital of Infectious Diseases in Bucharest
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Optic Nerve Sheath Diameter | Daily during the first week of hospitalisation
  The diameter of the optic nerve sheath measured ultrasonographically using a standardised method, 6mm from the surface of the retina

SECONDARY OUTCOMES:
C-reactive protein | Day 1, day 3 and day 7
  Measurement of systemic C-reactive protein (CRP) levels, as marker of systemic inflammation
Neuron-specific Enolase | Day 1, day 3 and day 7
  Measurement of neuron-specific enolase as a marker for brain cell death caused by CNS inflammation.
CSF examination | Day 1, day 3 and day 7
  Determining CSF immune cell count, CSF proteins, albumin, glucose, chloride and sodium, as well as bacterial or fungal cultures (where applicable).
Glasgow Coma Scale | Daily during the first week of hospitalisation
  Evaluation tool used to assess a person's level of consciousness after brain injury or illness, rating their eye, verbal, and motor responses for a total score ranging from 3 (deep unconsciousness) to 15 (fully alert).
Richmond Agitation-Sedation Scale | Daily during the first week of hospitalisation
  Ten-point clinical tool used in intensive care units to assess a patient's level of alertness, agitation, or sedation. Ranges from +4 (combative) to -5 (unarousable/comatose), 0 being alert and calm.
Middle Cerebral Artery Pulsatility Index | Daily during the first week of hospitalisation
  Transcranial Doppler ultrasound used to measure the middle cerebral artery (MCA) pulsatility index (PI).

CONTACTS AND LOCATIONS:
Overall Officials: Bogdan Pavel, MD, PhD, DESA, Principal Investigator — "Dr. Victor Babeș" Clinical Hospital for Infectious and Tropical Diseases
Locations (2):
- Romania (2):
  - Fundeni Clinical Institute, Bucharest, Bucharest
  - "Dr. Victor Babeș" Clinical Hospital for Infectious and Tropical Diseases, Bucharest, Bucharest

IPD SHARING:
Plan to Share IPD: Undecided